CLINICAL TRIAL: NCT02746523
Title: Later Life Cognitive Impairment, Proprioception, and Biomarkers in Former NHL Players Who Suffered Multiple Concussions
Brief Title: Effects of Multiple Concussions in Retired NHL Players
Acronym: NHL
Status: Terminated | Type: Observational
Why Stopped: Could not recruit enough subjects
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Assistant Professor, Ph. D., New York Institute of Technology
Other Study IDs: BHS-1170
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Cognitive Deficits; Proprioceptive Disorders
Keywords: NHL; Concussion; Biomarkers
MeSH Terms: conditions — Cognition Disorders; Somatosensory Disorders; Brain Concussion | interventions — Biomarkers; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, nasal swab, mouth swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case / Retired NHL Players: All interventions for this group are described below:
  Sensory Organization Test (SOT): Balance and proprioception test
  Connor's Adult ADHD Rating Scale (CAARS): A computer based questionnaire used to measure the presence of adult attention deficit hyperactivity disorder.
  Beck's Depression Inventory: A 21 question multiple choice self report measuring the severity of depression
  Patient Health Questionnaire 9 (PHQ-9): Self administered screening questionnaire for mental health disorders
  Montreal Cognitive Assessment (MoCA): A validated screening tool to assess cognitive mild impairment
  Blood/Urine/Saliva Biomarker analysis: These samples will be analyzed for relevant biomarkers
  Interventions: Other: Sensory Organization Test; Genetic: Biomarkers; Other: Conners' Adult ADHD Rating Scale (CAARS); Other: Depression Scale; Other: Cognitive Assessment
- Age Matched Controls: All interventions for this group are described below:
  Sensory Organization Test (SOT): Balance and proprioception test
  Connor's Adult ADHD Rating Scale (CAARS): A computer based questionnaire used to measure the presence of adult attention deficit hyperactivity disorder.
  Beck's Depression Inventory: A 21 question multiple choice self report measuring the severity of depression
  Patient Health Questionnaire 9 (PHQ-9): Self administered screening questionnaire for mental health disorders
  Montreal Cognitive Assessment (MoCA): A validated screening tool to assess cognitive mild impairment
  Blood/Urine/Saliva Biomarker analysis: These samples will be analyzed for relevant biomarkers
  Interventions: Other: Sensory Organization Test; Genetic: Biomarkers; Other: Conners' Adult ADHD Rating Scale (CAARS); Other: Depression Scale; Other: Cognitive Assessment

INTERVENTIONS:
Other: Sensory Organization Test — Balance and proprioception test
Genetic: Biomarkers — Blood, urine, and saliva biomarkers
Other: Conners' Adult ADHD Rating Scale (CAARS) — Adult ADHD rating scale
Other: Depression Scale — Becks Depression Inventory and Patient Health Questionnaire 9 (PHQ-9)
Other: Cognitive Assessment — Montreal Cognitive Assessment (MoCA)

SUMMARY:
To investigate long term affects of multiple concussions on the cognition, balance, proprioception, and biomarkers in retired National Hockey League players

DETAILED DESCRIPTION:
This research study will collect data for each subject in one single visit. During the visit the subject will be asked to consent to the study which is estimated to take approximately 10 minutes. A medical history will be obtained, taking approximately 15 minutes. Blood, urine, and cheek swabs will be collected for approximately 15 minutes. The PHQ-9, Becks Depression Inventory, Connors Adult ADHD Rating Scale (CAARS™), and Montreal Cognitive Assessment (MoCA) will be administered, these assessments combined are estimated to take 50 minutes. Lastly, patients will be asked to complete a Sensory Organization Test (SOT) which takes approximately 15 minutes. There are only licensed health professionals working on this project that will respect your privacy and conduct this trial following all HIPPA and clinical research guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Retired professional NHL player
* History or reported concussion and concussion like symptoms

Exclusion Criteria:

* Any neurological condition
* Non sport related head trauma

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retired NHL Players who suffered multiple concussions and age matched controls
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cognition assessed with the Montreal Cognitive Assessment Scale | 10 minutes
  Montreal Cognitive Assessment Scale

SECONDARY OUTCOMES:
Beck's Depression Inventory | 10 minutes
  A 21 question multiple choice self report inventory measuring the severity of depression
Adult Attention Deficit assessed with the Connors' Adult Attention Deficit Disorder Rating Scale | 10 minutes
  Connors' Adult Attention Deficit Disorder Rating Scale
Proprioception/Postural Stability assessed with the Sensory Organization Test | 15 minutes
  Sensory Organization Test
Human Interleukin-6 (IL-6) | 5 Minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed biomarkers Marker type: Inflammation
Patient Health Questionnaire 9 (PHQ-9) | 5 minutes
  Self administered screening and diagnostic questionnaire for mental health disorders
Interleukin 7 (IL-7) | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed biomarkers Marker Type: Inflammation
Human 8-hydroxy-2' -deoxyguanosine (8-OHdG) | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Oxidative stress on DNA
3-nitrotyrosine | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Oxidative stress on lipids
8-iso-Prostaglandin F2a | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: oxidative stress on lipids
Dityrosine | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Oxidative Stress on protein
Apolipoprotein E-4 | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Traumatic brain injury
Complement Component 3 B (C3b) | 5 minutes
  Blood (20 cc), Urine (40 cc), Saliva (5 cc): Total volume for all proposed Marker Type: Complement system
MicroRNA miR132 | 5 minutes
  Blood (20 cc), Urine (40 cc), Saliva (5 cc) Total volume for all proposed Marker Type: MicroRNA
MicroRNA miR183 | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: MicroRNA
S-100B Calcium binding protein | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Blood brain barrier damage
Brain derived neurotrophic factor (BDNF) | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Inflammation
Amyloid beta 40 | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Neurodegeneration
Total Tau Protein (tTAU) | 5 minutes
  Blood (20 cc), Urine (40 cc): Total volume for all proposed Marker Type: Traumatic brain injury
Eco-Rna Species | 5 minutes
  Blood (20 cc), Urine (40 cc),Saliva (5 cc): Total volume for all proposed Marker Type: Exo-RNA

CONTACTS AND LOCATIONS:
Overall Officials: Brian Harper, MD, Study Chair — NYIT-COM
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participants data will not be shared with individuals